CLINICAL TRIAL: NCT02213666
Title: Comparison of Intracardiac Echocardiography and Transesophageal Echocardiography for Imaging of the Left Atrial Appendage and Right Atrial Appendage in Patients With Atrial Fibrillation
Brief Title: Comparison of Intracardiac Echocardiography and Transesophageal Echocardiography
Acronym: ICE-TEE
Status: Completed | Type: Observational
Sponsor: Elad Anter (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Elad Anter, Attending Physician, Cardiac Electrophysiology, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Other Study IDs: 2011P000387
Record Dates: First submitted 2014-07-15; First posted 2014-08-11 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Atrial Fibrillation; Atrial Flutter
Keywords: Atrial fibrillation ablation; Intracardiac echocardiography; Thrombus; Left atrial appendage; Right atrial appendage
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Thrombosis | interventions — Cardiac Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intracardiac and Transesophageal Echocardiography: Imaging of the right atrial appendage and left atrial appendage with ICE and TEE
  Interventions: Device: Intracardiac Imaging

INTERVENTIONS:
Device: Intracardiac Imaging — Imaging of the RAA and LAA with ICE and assessment of thrombus.
  Other Names: Siemens AcuNav 8 French Phased Array Intracardiac Ultrasound Catheter

SUMMARY:
The presence of intracardiac thrombi and their propensity for systemic embolism is a major concern in patients with atrial fibrillation (AF) and atrial flutter (AFL) undergoing cardioversion and ablation procedures. Transesophageal echocardiography (TEE) is the clinical gold standard imaging modality for visualization of the right atrial appendage (RAA) and left atrial appendage (LAA) for detection of thrombi as well as risk factors associated with thrombus formation, including spontaneous echo contrast and low LAA velocity. However, TEE is a moderately invasive procedure that incurs additional risk, cost, and patient discomfort. In addition, thrombus detection via TEE may be ambiguous, and another tool capable of confirming uncertain TEE findings is desirable. This is particularly crucial in cases when adequate LAA imaging cannot be acquired or if TEE is clinically contraindicated, requiring alternative imaging modalities that can visualize these structures.

Phased-array intracardiac echocardiography (ICE) provides high-imaging resolution and is routinely used during atrial fibrillation (AF) ablation procedures for transseptal puncture and periprocedural catheter visualization. A majority of imaging acquired during AF ablation is performed with the ICE catheter in the right atrium (RA). However, these standard views are often unable to provide sufficient visualization of the LAA structure due to the relatively long distance between the ICE catheter and LAA.

Placement of the ICE catheter in the pulmonary artery (PA) provides improved visualization of the LAA over other locations by reducing the anatomic distance between the imaging catheter and structure of interest. Recent retrospective studies have confirmed improved assessment of the LAA with ICE imaging from the PA and equivocal sensitivity and specificity when compared with TEE for evaluation of LAA thrombus. However, these studies did not systematically evaluate the presence of SEC, flow velocity, the LAA dimensions, or the RAA.

Although these studies support the use of ICE imaging from the PA to clarify or confirm TEE findings, a prospective and blinded study evaluating both the LAA and RAA in its entirety is required. We hypothesize that this prospective and blinded study will confirm ICE as non-inferior to TEE in the assessment of LAA and RAA structure and for the detection of thrombi.

DETAILED DESCRIPTION:
Transesophageal echocardiography (TEE) is the clinical standard for diagnosis of left atrial appendage (LAA) and right atrial appendage (RAA) thrombi before cardioversion or instrumentation of the left atrium during ablation proce- dures.1-5 Occasionally, TEE cannot be performed because of anatomic limitations requiring an alternative imaging strategy to exclude LAA thrombi. Phased-array intracardiac echocardiography (ICE) is routinely used during atrial fibrillation (AF) ablation procedures to guide transseptal puncture and detect complications. The standard position of the transducer is in the right atrium (RA). This allows adequate visualization of the interatrial septum and body of the left atrium (LA) but not of the LAA because of significant physical distance from the transducer. Imaging of the LAA from closer anatomic structures such as the right ventricular outflow tract (RVOT) and pulmonary artery (PA) can improve visualization of the LAA. If ICE provided imaging of the LAA comparable to TEE with a good safety profile, it could potentially serve as an alternative to TEE in patients undergoing catheter ablation. Such an approach could reduce risk, cost, and patient discomfort associated with TEE combined with ICE. In this prospective blinded study, we sought to directly compare the sensitivity and specificity of TEE with ICE for detection of LAA and RAA anatomy and thrombus in patients with atrial tachyarrhythmias undergoing catheter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand and critically review the informed consent.
* Patients presenting for an AF and/or AFL ablation procedure who have clinical indication for TEE and ICE.

Exclusion Criteria:

* Patients in whom placement of an ICE catheter for adequate atrial visualization is technically not feasible.
* Patients requiring urgent cardioversion.
* Patients with a contraindication for TEE
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with drug-refractory, symptomatic, paroxysmal or persistent atrial fibrillation or atrial flutter requiring a clinical indicated ablation procedure.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elad Anter, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Cory M Tschabrunn, CEPS, Study Director — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were interviewed in the pre-procedure room on the day of the planned procedure after consenting for the planned clinical procedure. A Co-Investigator introduced and discussed the study with the patient in detail, provided the consent form to review and addressed any questions.
Groups:
- Intracardiac and Transesophageal Echocardiography: The study sample includes patients referred for a clinically indicated ablation procedure of atrial fibrillation or atrial flutter.
Period: Overall Study
Arm/Group | Intracardiac and Transesophageal Echocardiography
Started | 72
Completed | 71
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Patients enrolled into study that underwent ICE and TEE imaging.
Groups:
- Enrolled Patients: The study sample includes patients referred for a clinically indicated ablation procedure of atrial fibrillation or atrial flutter.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Intracardiac and Transesophageal Echo Results
Description: The right atrial appendage (RAA) and left atrial appendage (LAA) will be assessed for the presence or absence of intracardiac thrombi with the Siemens AcuNav Ultrasound catheter. This is also performed with the standard of care modality, transesophageal echocardiography (TEE) with both operators blinded to the opposing imaging modality. The presence of LAA thrombi requires cancellation of the clinical procedure. After a determination has been made by both operators regarding the presence or absence of thrombi will investigators be unblinded to the opposing imaging modality result. If intracardiac thrombi was detected, the procedure was cancelled according to standard clinical guidelines and practice. There is no follow-up data collected. Participants were followed during enrollment and the clinical ablation procedure which is an average of a 6 hour period.
Time Frame: Time of Clinical Procedure Only (Average 6 hours)
Measure: Number; unit: participants
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 71
participants
  Intracardiac Echo Completed | 71
  TEE Completed | 69
  Total Cases of Definite Thrombi Identified | 4
  TEE Diagnostic in Identification of Thrombi | 1
  ICE Diagnostic in Identification of Thrombi | 4

ADVERSE EVENTS:
Time Frame: During enrollment, the clinical ablation procedure, while in the hospital.
Description: All patients were screened for any complications at the conclusion of the clinical procedure (average of 6 hour period).
Arm/Group | Enrolled Patients
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 2/71
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled Patients (N=71)
Oropharyngeal bleeding from TEE (Surgical and medical procedures) | 2 (2) — 2 patients developed oropharyngeal bleeding from the TEE probe - this is a known complication associated with TEE imaging and not associated with participation in the study. This resolved spontaneously without further consequence or intervention.

LIMITATIONS AND CAVEATS:
This study compared TEE and ICE for visualization of the LAA and RAA in a specific patient population with nonvalvular AF treated with chronic anti-coagulation. The utility of ICE in other patient populations has not been examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No